CLINICAL TRIAL: NCT04993001
Title: Impact of an Open Lung Extubation Strategy on Postoperative Pulmonary Complications Compared to a Conventional Extubation Strategy: a Pilot Study
Brief Title: Impact of an Open Lung Extubation Strategy on Postoperative Pulmonary Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21.126
Record Dates: First submitted 2021-07-26; First posted 2021-08-06 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia; Pulmonary Atelectasis; Complication of Anesthesia
Keywords: Open lung extubation strategy; Postoperative pulmonary complications
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Pilot, single-center, randomized, triple-blind controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergence from general anesthesia with an open lung extubation strategy (Active Comparator)
  Interventions: Other: Open lung extubation
- Emergence from general anesthesia with a conventional extubation strategy (Placebo Comparator)
  Interventions: Other: Conventional extubation

INTERVENTIONS:
Other: Open lung extubation — Before starting emergence from anesthesia, the patient will be transferred to their hospital bed or stretcher and seated at 30 degrees. Secretions from the patients' oropharynx will be suctioned. To prevent the patient from coughing, the anesthetic gas or intravenous agent will be stopped after the transfer and suction procedure are completed. The FiO2 will be maintained at the same level or increased to 50% (minimum FiO2) with a fresh gas flow rate greater than or equal to 10 L.min-1. The ventilation mode will be changed to pressure support. The level of pressure support will be modified by the anesthesiologist to generate the same volumes as with controlled ventilation. The PEEP will be maintained at the same level. The minimum respiratory rate will be reduced by 4 min-1. The inspiratory flow for triggering will be 2 L.min-1.
  Arms: Emergence from general anesthesia with an open lung extubation strategy
Other: Conventional extubation — Before starting emergence from anesthesia, the patient will be transferred to his hospital bed or stretcher and kept in the supine position. Secretions from the patients' oropharynx will be suctioned. To prevent the patient from coughing, the anesthetic gas or intravenous agent will be stopped after the transfer and suction procedure are completed. The FiO2 will be increased to 100% with a fresh gas flow rate greater than or equal to 10 L.min-1. The ventilator will be stopped with the APL valve open to atmosphere. The patient will be manually ventilated with the reservoir bag until spontaneous ventilation resumes. Then, the patient may be manually assisted if the treating anesthesiologist deems it necessary.
  Arms: Emergence from general anesthesia with a conventional extubation strategy

SUMMARY:
Perioperative respiratory complications are a major source of morbidity and mortality. Postoperative atelectasis plays a central role in their development. Protective "open lung" mechanical ventilation aims to minimize the occurrence of atelectasis during the perioperative period. Randomized controlled studies have been performed comparing various "open lung" ventilation protocols, but these studies report varying and conflicting effects. The interpretation of these studies is complicated by the absence of imagery supporting the pulmonary impact associated with the use of different ventilation strategies. Imaging studies suggest that the gain in pulmonary gas content in "open lung" ventilation regimens disappears within minutes after the extubation. Thus, the potential benefits of open-lung ventilation appear to be lost if, at the time of extubation, no measures are used to keep the lungs well aerated. Recent expert recommendations on good mechanical ventilation practices in the operating room conclude that there is actually no quality study on extubation.

Extubation is a very common practice for anesthesiologists as part of their daily clinical practice. It is therefore imperative to generate evidence on good clinical practice during anesthetic emergence in order to potentially identify an effective extubation strategy to reduce postoperative pulmonary complications.

DETAILED DESCRIPTION:
The aim of this study is to establish the feasibility of a multicenter randomized controlled clinical trial comparing two clinical strategies called "open lung" and "conventional" during extubation. The investigators also aim to estimate the rates of postoperative pulmonary complications in the two intervention groups and verify the hypothesis that the "open lung" extubation strategy improves postoperative lung aeration as measured by the quantitative Lung Ultrasound Score compared to a conventional extubation strategy.

Methods

A pilot, prospective, randomized and controlled triple-blind study. Sixty-nine patients scheduled to undergo elective surgery at the CHUM and at moderate or high risk of postoperative pulmonary complications according to the ARISCAT score will be recruited. Following the administration of standardized mechanical ventilation and after obtaining consent, participants will be randomly assigned to two groups: Intervention group, "open lung" extubation strategy and Control group, "conventional" extubation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age requiring elective surgery under general anesthesia and hospitalization.
* Patients with a moderate or high risk of postoperative pulmonary complication according to the ARISCAT score (score of 26 or more)

Exclusion Criteria:

* Expected or known difficult intubation according to the treating anesthesiologist
* Postoperative mechanical ventilation (planned or unplanned)
* Neuromuscular disease
* Intrathoracic surgery
* Respiratory failure, sepsis or mechanical ventilation in the month preceding anesthesia
* Pregnancy
* Patient refusal
* Ultrasound sub-study:

  * Body mass index greater than 40 kg.m-2
  * Extensive postoperative chest dressings
* Clinician's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Protocol adherence rate | At the end of the surgery
  During emergence from general anesthesia, a research assistant will observe the adherence to the protocol. The adherence rate will be defined as the number of extubations performed according to the protocol and the patient assigned group divided by the total number of awakenings. In the event of a breach of the protocol, the specific elements that led to the deviation will be noted as well as the reasons given by the treating anesthesiologist to justify it.

SECONDARY OUTCOMES:
Number of eligible patients per week | Through study completion, an average of 1 year
Rate of consent to participate in the protocol | Through study completion, an average of 1 year
Rate of missing values | Through study completion, an average of 1 year

OTHER OUTCOMES:
Estimated baseline rates of postoperative respiratory complications in the two intervention groups | 7 days following the patient enters the recovery room
  Postoperative pulmonary complications will be defined using the definition recommended by the StEP group. These will be compiled from the patient's arrival in the recovery room until the 7th postoperative day or, if earlier, until discharge from hospital. Adjudication of complications will be performed by 2 investigators blinded to the treatment group. Any disagreement will be resolved by discussion between the two reviewers.
Comparison of pulmonary aeration using the qLUS score in the two intervention groups | 15 minutes after the patient enters the recovery room
  A lung ultrasound will be performed on each patient during pre-emergence preparations and 15 minutes after the patient arrives in the recovery room. The quantitative Lung Ultrasound Score will be calculated for each ultrasound examination. The physician performing the ultrasound examinations will be kept blind from the intervention group.
Re-intubation rate in the operating room | At the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girard J, Zaouter C, Moore A, Carrier FM, Girard M. Effects of an open lung extubation strategy compared with a conventional extubation strategy on postoperative pulmonary complications after general anesthesia: a single-centre pilot randomized controlled trial. Can J Anaesth. 2023 Oct;70(10):1648-1659. doi: 10.1007/s12630-023-02533-z. Epub 2023 Jul 27. PMID 37498442